CLINICAL TRIAL: NCT06710652
Title: Efficacy and Safety of Transcranial Magnetic Stimulation in Treatment of Insomnia with Subjective Cognitive Decline: a Randomized Controlled Trail
Brief Title: Efficacy and Safety of Transcranial Magnetic Stimulation in Treatment of Insomnia with Subjective Cognitive Decline
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS-insomnia
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Insomnia Chronic; Subjective Cognitive Decline (SCD)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS (Experimental)
  Interventions: Device: rTMS
- sham rTMS (Sham Comparator)
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: rTMS — Stimulation coil Cool-B65 A CO, located right lingual gyrus, stimulation frequency 1Hz, stimulation intensity 80% of motor threshold, number of stimuli 3 pulses/train, train interval 1s, 500 trains in total, 1500 total stimulation pulses, total stimulation time 20 min, treatment application once a day, continuous application for two weeks, 5 days a week.
  Arms: rTMS
Device: Sham Comparator — Stimulation coil Cool-B65 P CO, located right lingual gyrus, stimulation frequency 1Hz, stimulation intensity 80% of motor threshold, number of stimuli 3 pulses/train, train interval 1s, 500 trains in total, 1500 total stimulation pulses, total stimulation time 20 min, treatment application once a day, continuous application for two weeks, 5 days a week.
  Arms: sham rTMS

SUMMARY:
Insomnia is the most common form of sleep disorder, and subjective cognitive decline (SCD) in patients with insomnia may be an ultra-early manifestation of AD. Repetitive transcranial magnetic stimulation (rTMS) has emerged as a promising tool for the treatment of insomnia by modulating neural excitability and inducing plasticity. However, there is a lack of studies on rTMS treatment of cognitive impairment associated with insomnia. The efficacy and safety of rTMS for cognitive impairment in insomnia patients with SCD will be assessed by a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 30-80 years old; (2) Diagnostic criteria for insomnia: DSM-V and ICSD-3; (3) Subjective cognitive decline. (4) Regular use of non-benzodiazepines for insomnia.

Exclusion Criteria:

* (1) Refuse participants; (2) Presence of cognitive dysfunction; (3) Combined with other diseases other than central nervous system non-neurodegenerative diseases; (4) Use drugs that may affect cognition, degree of awakening and sleep quality due to other diseases; (5) Contraindications to rTMS treatment: (6) Severe complications and immune diseases; (7) Inability to cooperate; (8) Pregnancy or lactation.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline SCD-Q9 to 2 weeks | Baseline vs 2 weeks after treatment
  9-item Subjective Cognitive Decline Questionnaire (SCD-Q9)
Change from baseline MMSE to 2 weeks | Baseline vs 2 weeks after treatment
  Mini-Mental State Examination (MMSE)

SECONDARY OUTCOMES:
Change from baseline MoCA scores to 2 weeks | Baseline vs 2 weeks after treatment
  Montreal Cognitive Assessment (MoCA)
Change from baseline CDR to 2 weeks | Baseline vs 2 weeks after treatment
  Clinical Dementia Rating (CDR)
Change from baseline RAVLT to 2 weeks | Baseline vs 2 weeks after treatment
  Rey Auditory Verbal Learning Test (RAVLT)
Change from baseline HAMA to 2 weeks | Baseline vs 2 weeks after treatment
  Human Anti-Murine Antibodies (HAMA)
Change from baseline HAMD to 2 weeks | Baseline vs 2 weeks after treatment
  Hamilton Rating Scale for Depression (HAMD)
Change from baseline NPI to 2 weeks | Baseline vs 2 weeks after treatment
  Neuropsychiatric Inventory (NPI)
Change from baseline CDS to 2 weeks | Baseline vs 2 weeks after treatment
  Coding Digit Symbol subtest (CDS)
Change from baseline DDS to 2 weeks | Baseline vs 2 weeks after treatment
  Direct Digit Span subtest (DDS)
Change from baseline inflammatory factors and neuropathological markers to 2 weeks | Baseline vs 2 weeks after treatment
  Aβ, tau, GFAP, α-Synuclein, NFL, VEGF, AQP4, RNA sequencing, pre.Caspase1, cl.Caspase1, pre.IL-1β, cl.IL-1β, IL-18, GSDMD, ASC, NLRP1, Iba-1, GFAP, NeuN, CD86, CD206, iNOS, Arg1, TLR4, TLR2, MyD88, NFκB, tau, p-NFκB, NLRP3, β-actin, ect.
Change from baseline PAF to 2 weeks | Baseline vs 2 weeks after treatment
  The alpha-peak frequency (PAF) is the frequency with the highest power within the alpha-band.
Change from baseline structural imaging indicators to 2 weeks | Baseline vs 2 weeks after treatment
  The intra-cellular compartment (Vic) of the Neurite Orientation Dispersion and Density Imaging (NODDI) model represents diffusion within the axons and cells.And NODDI models the dispersion of axonal fibers with the use of an Orientation Dispersion Index (ODI).
Change from baseline adverse events to 2 weeks | Baseline vs 2 weeks after treatment
  Headache, tinnitus, pure tone hearing disorder, ect.
Change from baseline TMS-EEG to 2 weeks | Baseline vs 2 weeks after treatment
  Concurrent transcranial magnetic stimulation and electroencephalography (TMS-EEG)

IPD SHARING:
Plan to Share IPD: No